CLINICAL TRIAL: NCT04965701
Title: First Line Osimertinib in the Real World: an Inter-regional Prospective Study: FLOWER
Brief Title: First Line Osimertinib in the Real World: an Inter-regional Prospective Study
Acronym: FLOWER
Status: Completed | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IOV-2020-FLOWER
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: EGF-R Positive Non-Small Cell Lung Cancer
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Untreated EGFR-mutant advanced non-small-cell lung cancer patients
  Interventions: Drug: Osimertinib 80 MG

INTERVENTIONS:
Drug: Osimertinib 80 MG — Osimertinib is administered according to clinical practice at the recommended dose of 80 mg, orally, once a day.

SUMMARY:
This study (FLOWER) will investigate effectiveness, safety, progression patterns and clinical management of untreated advanced NSCLC patients receiving fist-line osimertinib in the real-world.

DETAILED DESCRIPTION:
FLOWER is a real-world, prospective, observational study enrolling patients with histological and/or cytological diagnosis of EGFR-mutant aNSCLC, receiving first-line treatment with the third-generation EGFR-TKI, osimertinib. All the patients received osimertinib at the recommended dose of 80 mg, orally, once a day. Dosing interruptions or reductions required, based on individual tolerability, were managed according to clinical practice in compliance with label indications.

The FLOWER study aims at evaluating effectiveness, safety, progression pattern and clinical management of untreated EGFR-mutant aNSCLC patients in the real-world.

ELIGIBILITY:
Inclusion Criteria:

* histological confirmed diagnosis of NSCLC and EGFR mutation in exon 18-21;
* locally advanced inoperable or metastatic disease (stage III and IV according to 8th edition of the TNM classification for lung cancer);
* first line treatment with the third generation EGFR TKI, osimertinib;
* age >18 years
* written informed consent

Exclusion Criteria:

Patients who receive study drugs in clinical trials will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include histologically confirmed advanced/metastatic NSCLC patients with sensitizing alteration of EGFR receiving osimertinib treatment in first-line setting.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Median time to discontinuation (mTTD) | The primary analysis of mTTD will occur when all patients have had the opportunity to be treated for 6 months
  To evaluate the effectiveness of osimertinib in the real-world
Rate of treatment related adverse events (AEs) | The primary analysis of safety will occur when all patients have had the opportunity to be treated for 6 months
  to evaluate safety of patients treated with osimertinib in the real-world
Rate of dose reduction and temporary or definitive treatment interruption due to AE | The primary analysis of safety will occur when all patients have had the opportunity to be treated for 6 months
  to evaluate safety of patients treated with osimertinib in the real-world

SECONDARY OUTCOMES:
Median overall survival (mOS) | The primary analysis of mOS will occur when all patients have had the opportunity to be treated for 6 months
  To evaluate the effectiveness of osimertinib in the real-world
Median progression free survival (mPFS) | The primary analysis of mPFS will occur when all patients have had the opportunity to be treated for 6 months
  To evaluate the effectiveness of osimertinib in the real-world
Overall response rate | The primary analysis of ORR will occur when all patients have had the opportunity to be treated for 6 months
  To evaluate the effectiveness of osimertinib in the real-world
Progression pattern | The primary analysis of progression patterns will occur when all patients have had the opportunity to be treated for 6 months
  To evaluate the pattern of progression to first-line osimertinib in the real-world

OTHER OUTCOMES:
Diagnostic-therapeutic pathway of patients included in the study | The primary analysis of diagnostic-therapeutic pathways will occur when all patients have had the opportunity to be treated for 6 months
  To describe the diagnostic-therapeutic pathway of patients included in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto, Padua, Italy

IPD SHARING:
Plan to Share IPD: No